CLINICAL TRIAL: NCT06592300
Title: An Open Label, Balanced, Randomized, Two-sequence, Two-treatment, Four -Period, Single Oral Dose, Fully Replicate,Bioequivalence Study in Normal, Healthy, Adult, Human Subjects Under Fed Condition.
Brief Title: Bioequivalence Study of Two Products of Tenofovir Alafenamide 25 mg Film Tablet in Healthy, Adult, Human Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Humanis Saglık Anonim Sirketi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 0030-24
Record Dates: First submitted 2024-09-09; First posted 2024-09-19 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2024-09

CONDITIONS: Chronic Hepatitis B in Adults and Paediatric Patients
MeSH Terms: interventions — tenofovir alafenamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tenofovir Alafenamide Film Tablet (Experimental): Tenofovir Alafenamide 25 mg Film Tablet
  Interventions: Drug: Tenofovir Alafenamide Film coated Tablet; Drug: Vemlidy® film-coated tablets
- Vemlidy® film-coated tablets (Active Comparator): Vemlidy® 25 mg film-coated tablets
  Interventions: Drug: Tenofovir Alafenamide Film coated Tablet; Drug: Vemlidy® film-coated tablets

INTERVENTIONS:
Drug: Tenofovir Alafenamide Film coated Tablet — The administration was performed in the morning, 30 minutes after a high-fat, high-calorie vegetarian breakfast was served following an overnight fast of at least 10 hours.
Drug: Vemlidy® film-coated tablets — The administration was performed in the morning, 30 minutes after a high-fat, high-calorie vegetarian breakfast was served following an overnight fast of at least 10 hours.

SUMMARY:
To compare the bioavailability and characterize the pharmacokinetic profile of the sponsor's test product relative to that of reference product after single oral dose, fully replicate, bioequivalence study in normal, healthy, adult, human subjects under fed condition.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoker, Normal, healthy, adult, human, subjects between 18 and 45 years of age (both inclusive).
* Having a Body Mass Index (BMI) between 18.5 to 30.0 (both inclusive), calculated as weight in kg/height in m2.
* Not having significant diseases or clinically significant abnormal findings during screening, medical history, clinical examination, laboratory evaluations, 12 lead ECG, and chest X-ray recordings (P/A view).
* Able to understand and comply with the study procedures, in the opinion of the investigator.
* Able to give voluntary written informed consent for participation in the trial.
* In case of female subjects:

  i. Surgically sterilized at least 6 months prior to study participation. Or If of child bearing potential 1s willing to use a suitable and effective double barrier contraceptive method or intra uterine device during the study.

And ii. Serum pregnancy test must be negative

Exclusion Criteria:

* Known hypersensitivity or idiosyncratic reaction to Tenofovir alafenamide or any of the excipients or any related drug.
* History or presence of any disease or condition which might compromise the haemopoietic, renal, hepatic, endocrine, pulmonary, central nervous, cardiovascular, immunological, dermatological, gastrointestinal or any other body system.
* Ingestion or Use of medication [prescribed & over the counter (OTC) medication including but not limited to herbal medicines, Oxcarbazepine ,Phenobarbital, Phenytoin, Itraconazole, Ketoconazole ,Rifampicin ,Rifapentine, Rifabutin, Tipranavir/ritonavir)] at any time from 14 days prior to dosing of period-I and any vaccine (including COVID-19 vaccine) within 14 days prior to dosing of period-I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Any history or presence of asthma (including aspirin induced asthma) or nasal polyp or NSAIDs induced urticaria.
* Consumption of grap_efruits or its products within a period of 72 hours prior to dosing of period-I.
* Smokers or who have smoked within last 06 months prior to start of the study.
* A recent history of harmful use of alcohol (less than 2 years), i.e. alcohol consumption of more than 14 standard drinks per week for men and more than 7 standard drinks per week for women (A standard drink is defined as 360 mL of beer or 150 mL of wine or 45 ml of 40% distilled spirits, such as rum, whisky, brandy etc) or consumption of alcohol or alcoholic products within 48 hours prior to dosing of period-I.
* The presence of clinically significant abnormal laboratory values during screening.
* Use of any recreational drugs or history of drug addiction or testing positive in pre-study drug scans.
* History or presence of seizure or psychiatric disorder.
* A history of difficulty with donating blood.
* Donation of blood (1 unit or 350 mL) within a period of 90 days prior to the first dose of study medication.
* Receipt of an investigational medicinal product or participation in a drug research study within a period of 90 days prior to the first dose of study medication**.

  ** If investigational medicinal product is received within 90 days where there is no blood loss except safety lab testing, subject can be included considering 10 half-lives duration of investigational medicinal product received.
* Difficulty in swallowing oral solid dosage form like capsule or tablet.
* A positive hepatitis screen including hepatitis B surface antigen and/or HCV ntibodies.
* A positive test result for HIV antibody (1 &/or 2).
* An unusual diet, for whatever reason (for example, fasting, high potassium or low sodium), for four weeks prior to receiving the study drug in period I. In any such case subject selection will be at the discretion of the Principal Investigator.
* Subject with rare Hereditary problems of galactose intolerance, total lactase deficiency or glucosegalactose malabsorption.
* Nursing mothers (for female subjects).

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2024-07-06 (Actual); Primary Completion 2024-08-02 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | 6 hours
  If the reference product intra-subject CV is less than or equal to 30% for Cmax, then the 90% confidence interval of the relative mean Cmax of the test to reference formulation for Ln-transformed data was to be within 80.00% to 125.00%.
AArea under the plasma concentration curve from administration to last observed concentration at time t (AUC0-t) | 6 hours
  The 90% confidence interval of the relative mean (Geometric mean) of the Test to reference formulation for Ln-transformed AUCt was to be within 80.00% to 125.00%

SECONDARY OUTCOMES:
Time until Cmax is reached (Tmax) | 6 hours
  Descriptive Statistics
Area under the plasma concentration curve extrapolated to infinite time (AUC0-∞) | 6 hours
  Descriptive Statistics

CONTACTS AND LOCATIONS:
Locations (1):
- Lambda Therapeutic Research Ltd., Ahmedabad, Gujarat, India